CLINICAL TRIAL: NCT02238431
Title: Down-regulated Hormonally Controlled Cycles for Vitrification-warmed Blastocyst Transfers: Reduces Time to Transfer and Cycle Cancellation
Brief Title: Down-regulated Hormonally Controlled Cycles for Vitrification-warmed Blastocyst Transfers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient uptake
Sponsor: Antalya IVF (Other)
Responsible Party: Principal Investigator, Kevin Coetzee, Scientific Advisor, Antalya IVF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lucrin depot FET cycle; FET cycle cancellation (Other: Antalya IVF)
Record Dates: First submitted 2014-09-05; First posted 2014-09-12 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy
Keywords: Lucrin depot,; frozen embryo transfer,; artificial cycle,; pregnancy,; cancellation
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lucrin depot, artificial cycle start (Experimental): intramuscular administration of Lucrin depot (half dose of 3.75mg) on the 5th day following oocyte retrieval
  Interventions: Drug: Lucrin depot
- OCP active, artificial cycle start (Active Comparator): to take active OCP tablets (1 per day) from the 10th day following oocyte retrieval for at least 21 days
  Interventions: Drug: OCP
- Natural, menstrual period (Experimental): to wait for the second bleed to commence the artificial FET cycle
  Interventions: Other: Natural

INTERVENTIONS:
Drug: Lucrin depot — scheduling the start of the artificial cycle and hormone down regulation during the artificial cycle
  Arms: Lucrin depot, artificial cycle start
Drug: OCP — to schedule the start of the artificial cycle
  Arms: OCP active, artificial cycle start
Other: Natural — to use the normal menstrual period to schedule treatment start
  Arms: Natural, menstrual period

SUMMARY:
Currently all patients that have freeze-all ICSI treatment cycles have the start of their FET cycle scheduled with the use of OCP. While an excellent pregnancy rate (75%) for the patients that have a blastocyst transfer has been maintained over time, 15% of started FET cycles are being cancelled because of premature luteinization, and the treatment (to transfer) takes approximately 89 days. The use of a Lucrin depot may reduce the number of cycles cancelled and reduce the treatment time to approximately 69 days. The use of no drugs and allowing the normal menstrual cycle to determine the time to start the FET cycle may suit some patients. Whether these benefits can be obtained while still maintaining the current FET pregnancy rate will be the main focus of the trial.

DETAILED DESCRIPTION:
The patients will undergo standard assisted conception procedures; controlled ovarian stimulation (COS), oocyte pickup procedure (OPU), ICSI, embryo culture, blastocyst vitrification and frozen embryo transfer. If sufficient (>2) viable blastocyst develop from the in vitro culture of their embryos, all viable blastocysts will be cryopreserved using a routine vitrification procedure. This is the eligible patient population. On the day the last blastocyst(s) are frozen the patients will be given a further opportunity to ask questions and if satisfied they will be asked to complete a trial consent. At this point patients will be randomized by numeric code and given a schedule and drug prescription for scheduling the start of their hormone supplemented frozen embryo transfer cycle. During the scheduling period the patients will follow the drug prescription provided . After the completion of their treatment - the transfer of one or two vitrified-warmed blastocyst - the patients from both groups will receive identical luteal support drug schedules and prescriptions. A blood test will be performed on the 15th day of progesterone supplementation, to determine the βhCG blood concentration. Currently at Antalya IVF, approximately 75% of patients who have blastocysts transferred in a frozen embryo transfer cycle have a positive biochemical pregnancy test, >29 international units per litre (IU/L) of human chorionic gonadotropin (βhCG). If pregnant, patients will continue using estrogen and progesterone supplementation for a further 8 weeks. At 7 weeks of gestation (5 weeks after embryo transfer ) the patients will receive a transvaginal ultrasound scan (TVUS) to check for pregnancy viability (fetal sac with cardiac activity). Thereafter the patients will have regular TVUS to follow fetal development. At 20 weeks of gestation a TVUS will be performed to confirm an ongoing pregnancy (normal fetal development).

All drug packs are delivered to the clinic by the pharmacy after receiving the prescription. A staff member will verify the code on the prescription with randomization code allocated to the patient. The pack will then be given to the patient after verbally confirming patient identity. The packs will also contain a drug use instruction sheet and a trial information sheet.

ELIGIBILITY:
Inclusion Criteria:

* If patients have >2 blastocysts vitrified

Exclusion Criteria:

* All patients not willing to participate in the study
* Patients with any known adverse reaction to one or the other of the drugs prescribed
* All patients that have no surviving blastocysts for transfer

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Cycle cancellation | On day 14 of estrogen supplementation
  blood progesterone concentration (>2nmol/L) as a measure of premature luteinization

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 20 weeks of gestation
  TVUS normal fetal development >20 weeks of gestation, in case of a pregnancy

OTHER OUTCOMES:
Pregnancy | 15 days after start the start of progesterone supplementation
  >29 IU/L βhCG on day 15 from the start of progesterone supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya IVF, Antalya, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Gelbaya TA, Nardo LG, Hunter HR, Fitzgerald CT, Horne G, Pease EE, Brison DR, Lieberman BA. Cryopreserved-thawed embryo transfer in natural or down-regulated hormonally controlled cycles: a retrospective study. Fertil Steril. 2006 Mar;85(3):603-9. doi: 10.1016/j.fertnstert.2005.09.015. PMID 16500326
- [Background] Hill MJ, Miller KA, Frattarelli JL. A GnRH agonist and exogenous hormone stimulation protocol has a higher live-birth rate than a natural endogenous hormone protocol for frozen-thawed blastocyst-stage embryo transfer cycles: an analysis of 1391 cycles. Fertil Steril. 2010 Feb;93(2):416-22. doi: 10.1016/j.fertnstert.2008.11.027. Epub 2009 Jan 26. PMID 19171338
- [Result] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515